CLINICAL TRIAL: NCT01491932
Title: An Open-label Treatment Study to Evaluate the Safety, Tolerability and Efficacy of AFQ056 in Parkinson's Patients With L-dopa Induced Dyskinesias
Brief Title: Open-label, Long-term Safety Extension Study of AFQ056 in Parkinson's Patients With L-dopa Induced Dyskinesias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAFQ056A2299; 2011-004378-27 (EudraCT Number)
Record Dates: First submitted 2011-12-01; First posted 2011-12-14 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2017-03

CONDITIONS: Dyskinesias; Parkinson Disease; Movement Disorders; Parkinsonian Disorders; Anti-Dyskinesia Agents
Keywords: Parkinson Disease; L-dopa; Levodopa; Dyskinesia
MeSH Terms: conditions — Dyskinesias; Parkinson Disease; Movement Disorders; Parkinsonian Disorders | interventions — mavoglurant

ARMS (1):
- AFQ056 (Experimental): Patients entering the study will be titrated to target dose of AFQ056 twice daily or the highest tolerated dose at weekly intervals.
  Interventions: Drug: AFQ056

INTERVENTIONS:
Drug: AFQ056 — AFQ056 will be supplied as oral capsules.

SUMMARY:
This study is to evaluate long-term safety, tolerability and efficacy for AFQ056 in patients who have completed an AFQ056A study in Parkinson's disease L-dopa induced dyskinesias (PD-LID).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed a previous AFQ056A study or are eligible as defined in the core study protocol
* Outpatients
* Patients who have a primary caregiver willing and able to assess the condition of the patient throughout the study in accordance with protocol requirements

Exclusion Criteria:

* Atypical or secondary form of Parkinson's disease
* History of surgical treatment for PD including deep brain stimulation
* Advanced, severe, or unstable disease (other than PD)
* History of malignancy
* Evidence of dementia
* Untreated/ineffectively treated mental disorders
* Treatment with certain prohibited medications
* Abnormal lab values or heart abnormalities
* Pregnant or nursing women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adverse events including serious adverse events | Monitored for the duration of the study (anticipated to be an average of 3 years)
  The occurrence of adverse events would be sought by non-directive questioning of the patient at each visit. Adverse events may also be detected when they are volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessment.
Severity of adverse events including serious adverse events | Monitored for the duration of the study (anticipated to be an average of 3 years)
  The occurrence and severity of adverse events would be sought by non-directive questioning of the patient at each visit. Adverse events may also be detected when they are volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessment.
Change in vital signs from baseline to Weeks 1, 2, 4, 8, 12, Months 6, 9, 12, every 6 months thereafter. | Assessed at Day -14 to -3, Day 1, Weeks 1, 2, 4, 8, 12, Months 6, 9, 12, every 6 months thereafter
  Pulse and blood pressure at each visit as indicated above. If a patient discontinues in between these visits, this will be assessed at the time of discontinuation.
Changes in hematology/blood chemistry and urinalysis laboratory evaluations from baseline to Weeks 4, 8, 12, Months 6, 9, 12, every 6 months thereafter | Assessed at Day -14 to -3, Day 1(only urinalysis and only done if abnormalities), Weeks 4, 8, 12, Months 6, 9, 12, every 6 months thereafter
  Standard hematology with differential, aPTT, PT/INR;, clinical chemistry consists of albumin, alkaline phosphatase, amylase, total bilirubin, calcium, cholesterol, creatinine, CK, γ-GT, glucose, lipase, lactate dehydrogenase, inorganic phosphorus, magnesium, potassium, total protein, AST, ALT, sodium, triglycerides, urea and uric acid, FSH, LH, oxytocin, prolactin, TBG, TSH, and T4; urinalysis (specific gravity, protein, glucose and blood) If a patient discontinues in between these visits, these will be assessed at the time of discontinuation.
Change in ECGs from baseline to Weeks 4, 8, 12, Months 6, 9, 12, every 6 months thereafter | Assessed at Day -14 to -3, Day 1, (repeated if abnormalities seen), Weeks 4, 8, 12, Months 6, 9, 12, every 6 months thereafter
  A standard 12-lead ECG will be performed. A central facility will be used for interpretation and analysis of the ECGs. If a patient discontinues in between these visits, this will be assessed at the time of discontinuation.
Change in Unified Parkinson's Disease Rating Scale (UPDRS) part III scores from baseline to Weeks 4, 8, 12, Months 6, 9, 12, every 6 months thereafter | Assessed at Day 1, Weeks 4, 8, 12, Months 6, 9, 12, every 6 months thereafter
  Part III of the UPDRS (items 18-31; total score 0-56), has been proven to be a reliable instrument in assessing the anti-parkinsonian effect in PD patients. This scale measures 14 items such as speech, facial expression, tremor, action or postural tremor, rigidity, finger taps, hand movement, alternating movement, leg agility, arising from a chair, posture, gait, postural stability, and bradykinesia. A higher score is indicative of worsening of symptoms. If a patient discontinues in between these visits, this will be assessed at the time of discontinuation.
Incidence of AEs related to an exacerbation of the underlying movement disorder Parkinson's disease | Monitored for the duration of the study (anticipated to be an average of 3 years)
  The occurrence of adverse events relating to the underlying movement disorder Parkinson's disease would be sought by non-directive questioning of the patient at each visit. Adverse events may also be detected when they are volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessment.

SECONDARY OUTCOMES:
Change in mAIMS (modified Abnormal Involuntary Movement Scale) total score from baseline to Weeks 1, 2, 4, 8, 12, Months 6, 9, 12, every 6 months thereafter. | Assessed at Day 1, Weeks 1, 2, 4, 8, 12, Months 6, 9, 12, every 6 months thereafter
  The AIMS is a scale for assessing dyskinesia. The modified version of this scale used in this study focuses on 6 different parts of the body and rates abnormal movements from 0 (absence of dyskinesia) to 4 (severe) (maximal score, 24). If a patient discontinues in between these visits, this will be assessed at the time of discontinuation.
Change in Revised Lang-Fahn Activities of Daily Living Dyskinesia Scale (LFADLDS) scores (patient and caregiver versions) from baseline to Weeks 4, 12, Months 6, 9, 12, every 6 months thereafter | Assessed at Day 1, Weeks 4, 12, Months 6, 9, 12, every 6 months thereafter
  The LFADLDS is a questionnaire asking the patient about the degree to which dyskinesia interferes with activities of daily living. The LFADLDS is modified from the ADL section of the UPRDS (part II). Specific definitions for severity rating codes (range, 0-4 for each task) will be provided for reproducibility of results. A higher score indicates more severe impairment. Two versions of the revised LFADLDS will be used in this study: a patient version and a caregiver version. If a patient discontinues in between these visits, this will be assessed at the time of discontinuation.
Change in score for items 32, 33, and 34 of Part IV of the UPDRS from baseline to Weeks 4, 8, 12, Months 6, 9, 12, every 6 months thereafter | Assessed at Day 1, Weeks 4, 8, 12, Months 6, 9, 12, every 6 months thereafter
  The UPDRS is a standardized instrument for measuring the disease state of PD patients.
  Question 32 assesses duration of dyskinesias expressed in percentage of the day . Question 33 makes a historical assessment of disability due to dyskinesia during the previous week (not disabling, mildly disabling, moderately disabling, severely disabling, completely disabling).
  Question 34 of part IV assesses how painful the dyskinesias are from 0 (no painful dyskinesias) to 4 (marked). If a patient discontinues in between these visits, this will be assessed at the time of discontinuation.
Change in Mini Mental State Exam (MMSE) score from baseline to Months 6, 12, every 6 months thereafter | Assessed at Day -14 to -3, Day 1 (only if not done in the respective core study), Months 6, 12, every 6 months thereafter
  The MMSE is a brief test of cognitive dysfunction consisting of five sections (orientation, registration, attention-calculation, recall, and language) administered by a health care professional. The MMSE results in total possible score of 30, with higher scores indicating better function. If a patient discontinues in between these visits, this will be assessed at the time of discontinuation.
Change in the Scales for outcomes in Parkinson's disease - Psychiatric Complications (SCOPA-PC) score from baseline to Weeks 4, 8, 12, Months 6, 9, 12, every 6 months thereafter | Assessed at Day 1, Weeks 4, 8, 12, Months 6, 9, 12, every 6 months thereafter
  The SCOPA-PC is an easily administered semi-structured, questionnaire developed for the assessment of psychiatric symptoms, including compulsive behavior, in Parkinson's disease patients administered by a clinician with input provided by patient and caregiver. The total SCOPA score ranges from 0-21, with higher scores reflecting more psychiatric complications. If a patient discontinues in between these visits, this will be assessed at the time of discontinuation.
Proportion of patients who have suicidal ideation and behavior as mapped to Columbia Classification Algorithm for Suicide assessment (C-CASA) using data from Columbia-Suicide Severity Rating Scale (C-SSRS) | Monitored for the duration of the study (anticipated to be an average of 3 years)
  The C-SSRS assesses suicidal ideation/behavior using a patient interview. The data is mapped to Columbia Classification Algorithm for Suicide assessment. The code and categories are: completed suicide, suicide attempt, preparatory actions toward imminent suicide behavior, suicidal ideation, self-injurious behavior without suicidal intent.
  The proportion of patients who are coded in the categories above, the proportion of patients with any suicidal behavior engaged in during the study, and the proportion of patients with suicidality will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (30):
- United States (3):
  - Novartis Investigative Site, Englewood, Colorado
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Austria (3):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, London, Ontario, Canada
- France (3):
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Pessac
- Germany (8):
  - Novartis Investigative Site, Beelitz-Heilstätten
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Westerstede/Oldenburg
- Hungary (2):
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Szeged
- Italy (3):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Bratislava, Slovakia
- Spain (5):
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Bern, Switzerland

REFERENCES:
- See also: Results from CAFQ056A2299 from the Novartis Clinical Trial Results website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12843